CLINICAL TRIAL: NCT06646211
Title: A Single-arm, Multicenter Phase Ⅱclinical Study Evaluating High-dose Methotrexate Combined with Thiotepa and Zanubrutinib in the Treatment of Newly Diagnosed Central Nervous System Diffuse Large B-cell Lymphoma (MTZ)
Brief Title: High-dose Methotrexate Combined with Thiotepa and Zanubrutinib in the Treatment of Newly Diagnosed PCNSL (MTZ)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huiqiang Huang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-503-01
Record Dates: First submitted 2024-10-12; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL); Non Hodgkin Lymphoma (NHL)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — zanubrutinib; Thiotepa; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant Group/Arm： Experimental: Methotrexate , Thiotepa and Zanubrutinib(MTZ) (Experimental)
  Interventions: Drug: Zanubrutinib , Thiotepa; Drug: Methotrexate , Thiotepa and Zanubrutinib; Drug: ASCT±Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib , Thiotepa — First 1-4 cycle
  Drug: Thiotepa
  * 40mg/m2，d1 each 21-day cycle from cycle 1 for up to 4 cycle Drug: Zanubrutinib
  * Zanubrutinib will be given at a dose of 160mg，bid，d1-d21
Drug: Methotrexate , Thiotepa and Zanubrutinib — Cycle 5 - 10 Drug: Methotrexate
  * Intravenous methotrexate at 3.5g/m2 for 6 hours will be given on day 1 each 21-day cycle 【Leucovorin Calcium (CF): 15mg/m², rescue begins 12 hours after the infusion of methotrexate (MTX) ends, administered every 6 hours until the MTX plasma concentration is ≤ 0.1 μmol·L-¹ at 48 hours; plasma concentration monitoring time points: 0, 6, 24, 48, 72 hours.】 Other Names: MTX Drug: Thiotepa
  * 40mg/m2，d1 each 21-day cycle from cycle 5 for up to 10 cycle Drug: Zanubrutinib Zanubrutinib will be given at a dose of 160mg，bid，d1-d21
Drug: ASCT±Zanubrutinib — Consolidation / maintenance treatment Patients who achieve a Complete Response (CR) or Partial Response (PR) after the ZT/ZMT treatment will enter consolidation/maintenance therapy.
  Patients age ≤65 years old will undergo Autologous Stem Cell Transplantation (ASCT, with a recommended conditioning regimen that includes Thiotepa), followed by 6 months of maintenance treatment with zanubrutinib.
  Patients age > 65 will receive 6 months of maintenance treatment with zanubrutinib.
  *The study permits the prophylactic use of Granulocyte Colony-Stimulating Factor (G-CSF). For detailed usage, please refer to the guidelines from the National Comprehensive Cancer Network (NCCN) or the Chinese Society of Clinical Oncology (CSCO)

SUMMARY:
This is a phase Ⅱ clinical study of Zanubrutinib(Z) in combination with methotrexate (M) and thiotepa(T) in treating newly diagnosed primary CNS lymphoma (PCNSL).

The purpose of the study is to test the efficacy and tolerability of a combination treatment of MTZ regimen in treating patients who have newly diagnosed PCNSL

DETAILED DESCRIPTION:
PCNSL is a rare extranodal aggressive lymphoma accounting for 4%- 6% of all extranodal lymphomas and 3%- 4% of brain tumors, with an overall low incidence rate. However, with the extension of life expectancy, the incidence of PCNSL has increased by 2-3 times in Western Europe and the United States over the past 20 years.

Conventional dose methotrexate (MTX) does not effectively cross the blood-brain barrier, and the treatment for newly diagnosed PCNSL is still based on high-dose methotrexate (HD-MTX) combined chemotherapy. In the early stages PCNSL, Batchelor et al. used an MTX dose of 8.0g/m², which could reach effective therapeutic concentrations in the cerebrospinal fluid (CSF). However, HD-MTX has significant nephrotoxicity, especially for elderly patients and those with renal insufficiency. In 2005, Khan et al. found that reducing the dose of MTX to 3.5g/m² could significantly reduce kidney toxicity. Although single-agent HD-MTX has some efficacy in treating PCNSL, the remission rate is still relatively low. High doses of cytarabine, dacarbazine, and thiotepa have a higher blood-brain barrier penetration rate, and these drugs combined with HD-MTX for treating PCNSL can further improve upon HD-MTX alone. The overall response rate (ORR) is approximately 60%-70%, the complete response (CR) rate is about 40%-50%, and the 5-year survival rate is around 30%. Neither the short-term efficacy nor the long-term survival is satisfactory.

Basic research has found that excessive activation of the BCR signaling pathway in PCNSL tumor tissue, and BTK inhibitors such as ibrutinib can effectively inhibit the BCR pathway to achieve therapeutic goals. A study used single agent ibrutinib to treat relapsed/refractory PCNSL, with an overall response rate (ORR) of 50%. Grommes et al. reported that ibrutinib combined with high-dose methotrexate (HD-MTX) with or without rituximab showed specific efficacy in treating relapsed/refractory PCNSL, with an ORR of 89% and a complete response (CR) rate of 67%. The efficacy was significantly higher than that of single-agent ibrutinib in treating relapsed/refractory PCNSL.

Based on these studies, we hypothesize that first-line treatment with BTK inhibitors combined with HD-MTX-based chemotherapy may further improve the efficacy of newly diagnosed PCNSL and prolong the duration of remission.However, as a first-generation BTK inhibitor, ibrutinib has a relatively high off-target effect, leading to increased drug resistance and adverse reaction rates. Zanubrutinib, as a new generation of BTK inhibitors, has shown more potent antitumor activity and lower adverse reactions than ibrutinib in head-to-head clinical studies. Previously, we conducted a phase II clinical study of ibrutinib combined with methotrexate and temozolomide in PCNSL, which showed that ibrutinib significantly improved patients' overall response rate and complete response rate. However, the duration of remission was relatively short. Therefore, this study uses the new generation of zanubrutinib and thiotepa, which have intense penetration into the central nervous system, aiming to improve patients' remission duration further.

At the same time, based on previous studies and clinical experience, elderly and patients with renal insufficiency have poor tolerance to methotrexate, often experiencing delayed MTX clearance and renal damage. The first four courses of this study removed methotrexate and only used the less toxic zanubrutiniba and thiotepa, providing a reference for future methotrexate-free treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Men and woman who are 18 to 70 years of age
2. Histologically documented PCNSL
3. ECOG performance status ≤ 2
4. Life expectancy of > 3 months
5. Imaging show at least one measurable lesion in the central nervous system.
6. Adequate bone marrow and organ function shown by:
7. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
8. Platelets ≥ 75 x 10^9/L and no platelet transfusion within the past 14 days
9. Hemoglobin (Hgb) ≥ 8 g/dL and no red blood cell (RBC) transfusion within the past 14 days
10. International Normalized Ratio (INR) ≤ 1.5 and PTT (aPTT) ≤ 1.5 times the upper limit of normal
11. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3×ULN
12. Serum bilirubin ≤ 1.5×ULN
13. Serum creatinine ≤ 2×ULN
14. Lipase ≤ 1.5 x LUN
15. Women of childbearing potential (WOCBP) and men must agree to use effective contraception when sexually active. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of medication; women who are pregnant or breastfeeding are not eligible to participate in this study. Women of childbearing potential: from the time of signing the Informed Consent Form (ICF) until 30 days after the study ends, sexually active men: from the time of signing the ICF until 90 days after the study ends, must use contraceptive measures.
16. Must be able to tolerate MRI/CT scans
17. Must be able to tolerate lumbar puncture and/or Ommaya tap

Exclusion Criteria:

1. Diagnosed with a malignant tumor other than PCNSL or has received treatment, except for the following cases:

   1. Received curative treatment and has no known active disease at least 3 years or more before screening for enrollment.
   2. Fully treated non-melanoma skin cancer or malignant lentigo, with no evidence of disease.
   3. Fully treated carcinoma in situ, with no evidence of disease currently.
2. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure (New York Heart Association > Class 2), unstable angina, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
3. Uncontrolled hypertension despite optimal medical management (per investigators assessment)
4. Patient has poorly controlled diabetes (per investigators assessment)
5. Patient is known to have an uncontrolled active systemic infection (>CTCAE grade 2) and recent infection requiring intravenous anti-infective treatment that was completed ≤14 days before the first dose of study drug
6. Cerebrovascular accident, deep vein thrombosis or pulmonary embolism within 3 months before the start of study treatment
7. Non-healing wound, ulcer or bone fracture in a short time
8. Known bleeding diathesis or hemophilia
9. Known history of infection with human immunodeficiency virus (HIV) or active stage of infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) . Active HBV infection must be confirmed by a positive test for HBV surface antigen or a positive test for hepatitis B core antibody with a positive determination of HBV DNA by polymerase chain reaction (PCR). For Hepatitis C virus (HCV), confirmation must be made by a positive test for HCV antibodies, unless the subject has been treated and has shown a sustained virological response. Note: Subjects with positive HCV antibodies who have been treated and have shown a sustained virological response (negative virus detection for at least 6 months after completing treatment) will not be excluded.
10. Patient underwent major systemic surgery ≤ 2 weeks prior to starting the trial treatment or who has not recovered from the side effects of such surgery
11. Unable to swallow capsules or disease significantly affecting gastrointestinal function
12. Life-threatening illness, medical conditions, or organ dysfunctions that may endanger the safety of the subject or put the study outcomes at risk.
13. Lactating or pregnant
14. Requires anticoagulation therapy with warfarin or equivalent vitamin K antagonists; requires treatment with potent CYP3A4/5 inhibitors.
15. Requires long-term use of dexamethasone ≥4mg/day or equivalent doses of corticosteroid formulations.
16. Requires treatment with immunosuppressive agents, including cyclosporine A, tacrolimus, and sirolimus. Patients must discontinue the use of immunosuppressive agents 28 days before receiving study medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) at the end of TZ / MTZ treatment, Investigator-Assessed | 12 month
  The overall response rate (ORR) including complete response (CR), and partial response (PR) according to the 2005 Response Criteria of the International Primary CNS Lymphoma Collaborative Group (IPCG)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) at the end of TZ treatment, Investigator-Assessed | 12 month
  The overall response rate (ORR) including complete response (CR), and partial response (PR) according to the 2005 Response Criteria of the International Primary CNS Lymphoma Collaborative Group (IPCG)
Duration of response（DOR） | 12 month
  Duration of response is defined as the time from the date of first occurrence of CR or PR to the date of the first documented PD or death due to any cause.
Progression-free survival (PFS) | 12 month
  defined as the time from treatment to disease progression or death from any cause.
Overall survival (OS) | 12 month
  defined as the time from treatment to death from any cause
Frequency and severity of adverse effects as defined by CTCAE version 5.0 | 12 month
  All subjects who received at least one dose of MTZ will be included in the safety analysis. Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No